CLINICAL TRIAL: NCT04052958
Title: DM-IMT - Controlled, Randomized, Three-arm Intervention Study on the Safety and Efficacy of Regular Respiratory Muscle Training in Patients With Myotonic Dystrophy Type 1
Acronym: DM-IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Benedikt Schoser, Neurologist, Senior Physician, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Version 1.2 (26. Juni 2019)
Record Dates: First submitted 2019-07-31; First posted 2019-08-12 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Strength Training (Active Comparator): Respiratory muscle strength training
  Interventions: Device: IMT - inspiratory muscle training
- Group 2: Endurance Training (Active Comparator): Respiratory muscle endurance training
  Interventions: Device: IMT - inspiratory muscle training
- Group 3: Control group (No Intervention): no training of respiratory muscles

INTERVENTIONS:
Device: IMT - inspiratory muscle training — respiratory strength or indurance training with respiratory therapy device
  Arms: Group 1: Strength Training; Group 2: Endurance Training

SUMMARY:
For some diseases, regular respiratory muscle training could delay the start of ventilation. For DM1, however, there are no clinically high-quality studies. Only a case description from the year 2006 showed a missing improvement of the symptoms after respiratory muscle training in one patient, accordingly there are no recommendations in this issue. Within the scope of this monocentric, three-arm, controlled intervention study, 45 patients with genetically confirmed type 1 myotonic dystrophy will be randomized in three groups of 15 patients each, age-, gender- and symptom-corrected by the MUSCULAR IMPAIRMENT RATING SCALE (MIRS). The DM1 patients will receive regular respiratory muscle training for a period of 9 months. The aim of this study is to evaluate the safety and effectiveness of regular inspiratory strength-breathing muscle training on 15 patients, the safety and effectiveness of regular inspiratory endurance respiratory muscle training on 15 patients, and the comparison to the natural course in 15 patients without training. Subsequently, we will provide treatment recommendations for respiratory training in DM1.

ELIGIBILITY:
Inclusion Criteria:

* the patient is willing and able to provide a signed informed consent form
* the patient is ≥ 18 years old
* the diagnosis of type 1 myotonic dystrophy has been confirmed by molecular genetics
* the patient is able and willing to perform pulmonary function tests (PFT) and blood sampling for capillary blood gas analysis (pO2, pCO2) throughout the study, to keep a diary and to complete questionnaires

Exclusion Criteria:

* the patient requires invasive ventilation (non-invasive ventilation is allowed).
* the patient uses non-invasive ventilation more than 16h/day.
* the patient participates in another clinical study that involves therapy.
* the patient cannot perform pulmonary function tests (PFT).
* the patient is diagnosed with central sleep apnea in polysomnography and not sufficiently treated with NIV ventilation.
* the patient is diagnosed with obstructive sleep apnea and not sufficiently treated with NIV ventilation.
* the patient cannot meet the requirements of the study, according to the investigator.
* the patient is unable to complete a 6-minute walking test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of recurrent inspiratory muscle training | nine months
  Intervention-related (serious) adverse events will be assessed as described in protocoll DM-IMT Version 1.2 (26/June/2019). For example a deterioration of > 15% of the FVC compared to the baseline measurements is defined as AE, as is the development of unusual myalgia of the respiratory muscles for more than 12 hours after the respiratory training. Detailed lists of patients experiencing adverse events or SAEs are reported. The severity of the adverse event is classified as mild, moderate or severe. Relationships of an AE to the training are categorized as unassociated, unlikely to be associated, possibly associated or associated. A separate list will be provided for patients who drop out of the study due to AEs. The frequency of adverse events leading to study termination is also summarized. Safety parameters also include lung function tests (PFT, including FVC, FEV1, MIP, MEP), physical examination, vital signs and clinical laboratory tests as required.

SECONDARY OUTCOMES:
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by MIP. | nine months
  The efficacy of the respiratory training is determined by the results of Maximal inspiratory pressure (MIP).
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by MIP. | nine months
  The efficacy of the respiratory training is determined by the results of Maximal inspiratory pressure (MIP).
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by MEP. | nine months
  The efficacy of the respiratory training is determined by the results of Maximal exspiratory pressure (MEP).
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by MEP. | nine months
  The efficacy of the respiratory training is determined by the results of Maximal exspiratory pressure (MEP).
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by FVC. | nine months
  The efficacy of the respiratory training is determined by the results of Forced Vital capacity (FVC).
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by FVC. | nine months
  The efficacy of the respiratory training is determined by the results of Forced Vital capacity (FVC).
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by FEV1. | nine months
  The efficacy of the respiratory training is determined by the results of Forced Expiratory Volume in 1 second (FEV1).
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by FEV1. | nine months
  The efficacy of the respiratory training is determined by the results of Forced Expiratory Volume in 1 second (FEV1).
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by pCO2. | nine months
  The efficacy of the respiratory training is determined by the results of pCO2 in capillary blood gas analysis.
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by pCO2. | nine months
  The efficacy of the respiratory training is determined by the results of pCO2 in capillary blood gas analysis.
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by pO2. | nine months
  The efficacy of the respiratory training is determined by the results of pO2 in capillary blood gas analysis.
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by pO2. | nine months
  The efficacy of the respiratory training is determined by the results of pO2 in capillary blood gas analysis.
Efficacy of recurrent inspiratory muscle strength training in 15 patients with type 1 myotonic dystrophy measured by pH. | nine months
  The efficacy of the respiratory training is determined by the results of pH in capillary blood gas analysis.
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by pH. | nine months
  The efficacy of the respiratory training is determined by the results of pH in capillary blood gas analysis.
Efficacy of recurrent inspiratory muscle endurance training in 15 patients with type 1 myotonic dystrophy measured by 6-minute-walk-test. | nine months
  The efficacy of the respiratory training is determined by the results of 6-minute-walk-test.
Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training compared to patients without training, measured by DM1-Activ. | nine months
  Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training will be measured by the result of DM1-ACTIV, a Rasch-built DM activity and participation scale for clinical use.
Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training compared to patients without training, measured by FDSS. | nine months
  Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training will be measured by the result of the FDSS - FATIGUE AND DAYTIME SLEEPINESS SCALE, a Rasch-built combined fatigue and daytime sleepiness scale specifically designed for patients with DM1.
Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training compared to patients without training, measured by the questionnaire Respicheck. | nine months
  Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training will be measured by the result of the RESPICHECK, a questionnaire on clinical symptoms of respiratory insufficiency.
Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training compared to patients without training, measured by a physical examination. | nine months
  Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training will be measured by the result of the physical examination.
Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training compared to patients without training, using the 6-minute-walk-test. | nine months
  Impact on the quality of life and muscular performance in DM1 patients after recurrent respiratory muscle training will be measured by the result of the 6-minute-walk-test.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wenninger, Dr.med., Principal Investigator — Neurologist
Locations (1):
- Friedrich-Baur-Institute, Dep. of Neurology Klinikum der Universitaet Muenchen Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT04052958/Prot_000.pdf